CLINICAL TRIAL: NCT00734838
Title: Optical Spectroscopy During Breast Cancer Surgery and Core Needle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00008003; NIH 5R01-CA-100559; W81XWH-09-1-0410 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Biopsy; Reduction mammoplasty
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core needle biopsy (Experimental): Patients needing a needle biopsy of a breast mass
  Interventions: Device: High Resolution Microendoscope
- Reduction mammoplasty (Placebo Comparator): Any patients scheduled for a reduction mammoplasty who would like to participate in a study to better understand breast cancer
  Interventions: Device: High Resolution Microendoscope

INTERVENTIONS:
Device: High Resolution Microendoscope — Using core biopsy and reduction mammoplasty tissue

SUMMARY:
The objective of the proposed research is to develop new diagnostic modalities based on optical spectroscopy (auto fluorescence, absorption, and scattering) for the diagnosis of breast cancer and test its performance as an adjunct to core needle biopsy. For the surgery part of the study, all patients scheduled to have a mastectomy or lumpectomy for the treatment of breast cancer will be asked if they would be willing to participate in this study. For the core needle biopsy part of the study, patients with a higher pre-probability of cancer (based on mammography) will be recruited to increase the number of patients with malignant lesions and enrolled in this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a needle biopsy of a breast mass

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2006-01; Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Optical signatures | Day of procedure (less than 10 minutes)
  The primary outcome of this study is the identification of the optical signatures of normal and cancerous tissue of the breast

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States